CLINICAL TRIAL: NCT05339737
Title: Validation of a New Multi-parameter Technology to Better Diagnose Pain in the Adult Intensive Care Population: The Nociception Level (NOL) Index
Brief Title: The Nociception Level (NOL) Index for Pain Assessment in the Adult Intensive Care Unit
Acronym: NOL-ICU
Status: Not yet recruiting | Type: Observational
Sponsor: McGill University (Other)
Collaborators: Jewish General Hospital (Other); Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Céline Gélinas, Full Professor, McGill University
Other Study IDs: MP-05-2022-2988; 168983 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2022-04-02; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Pain, Acute; Nociceptive Pain; Behavior; Critical Illness
MeSH Terms: conditions — Acute Pain; Nociceptive Pain; Behavior; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Nociception Level (NOL) Index — The NOL integrates multiple physiologic parameters that are captured through a finger probe with disposable sensor. These parameters include heart rate, heart rate variability, photoplethysmography pulse wave amplitude, skin conductance and temperature, and their time derivatives. All these parameters are analyzed simultaneously to provide the NOL index which can range from 0 to 100. Values >25 were found to be indicative of nociception and related-pain in the field of anesthesia. The investigators will use the Pain Monitoring Device-200 (PMD-200)TM, which offers the multi-parametric NOL index (0-100) (Medasense Biometrics Ltd., Ramat Gan, Israel), and was approved by Health Canada for clinical use in September 2017.

SUMMARY:
Assessing pain in the adult intensive care unit (ICU) is challenging because many patients are unable to communicate due to mechanical ventilation and sedation. Therefore, it is necessary to have alternative methods to assess pain in this vulnerable patient population. In this project, the use of a multi-parameter technology (i.e., the Nociception Level (NOL) index) will be tested for pain assessment in ICU adults. The NOL index is a value from 0 to 100 obtained by calculating different parameters (e.g., pulse, skin temperature) captured through a small probe placed on the patient's finger. The NOL was initially developed for assessing nociception, pain and analgesia in anesthetized patients undergoing surgery, and its use in the ICU is new. The NOL's use before, during and after standard care procedures known to be painful (e.g., tube or drain removal, suctioning of secretions through the endotracheal tube) and non-painful (e.g., cuff inflation to measure blood pressure, soft touch) in ICU adults. The NOL will be monitored in three groups: a) patients able to communicate so they can self-report their pain (gold standard criterion) and express behaviors, b) patients unable to communicate but express behaviors (reference criterion), and c) patients unable to communicate and to express behaviors. In the first group, patients will be asked to self-report their pain and procedural distress on a 0 to 10 scale. In the first and second group, patients will be assessed for pain using a standardized behavioral scale which will be completed by trained research staff. In the third group, only the NOL will be monitored. Analgesic and sedative medication administered to patients will also be documented from medical charts. The ability of the NOL to detect pain based on self-reports of pain and behavioral scores, and its ability to discriminate between painful and non-painful procedures will be examined. If found to be useful, the NOL could be used as an alternative measure of pain and improve its recognition and treatment in vulnerable ICU patients.

DETAILED DESCRIPTION:
Background: Assessing pain in adult intensive care units (ICU) is challenging because self-report is often non-feasible due to patients' critical care conditions, mechanical ventilation and/or sedation. The Critical-Care Pain Observation Tool (CPOT) is the reference standard alternative measure of pain, but patients must be capable of expressing behaviors. Therefore, these cannot be used in patients who are heavily sedated or unresponsive (e.g., in coma), and other pain assessment methods must be explored. Vital signs alone (e.g., heart rate, blood pressure) are not valid for ICU pain assessment with inter-individual variability being a major limiting factor. The newly developed Nociception Level (NOL) index (Medasense Biometrics Ltd., Ramat Gan, Israel) is a numeric value from 0 to 100 obtained from simultaneous different parameters including heart rate, heart rate variability, photoplethysmography pulse wave amplitude, skin conductance level, number of skin conductance fluctuations, skin temperature, and their time derivatives. A NOL value>25 would indicate nociception and related pain in the field of anesthesia. The NOL could adequately classify nociceptive versus non-nociceptive stimuli with an area under the curve (AUC) >0.90 in anesthetized patients. The use of the NOL in the ICU is new. The investigators completed pilot work showing feasibility and promising validity results of the NOL for the detection of self-reported pain intensity and CPOT scores as reference criteria during chest tube removal and endotracheal suctioning in medical and surgical ICU patients.

The goal of this study is to validate the NOL index for the assessment of nociception and related pain in the ICU. Specific objectives are to examine the NOL's ability to:

1. detect pain in patients able to self-report and in non-communicative patients able to exhibit behavioral responses (i.e., criterion validation);
2. correlate with the patients' self-reports of procedural pain distress during nociceptive procedures (i.e., convergent validation); and
3. discriminate between non-nociceptive and nociceptive procedures as well as before and after the administration of a breakthrough dose of an opioid (i.e., discriminative validation).

As a complementary objective, feasibility and clinical utility of the NOL's use will be described from the ICU nurses' perspective.

Methods: A prospective cohort observational design will be used in two medical-surgical ICUs in Montreal where the research team has developed the expertise in the NOL's use. Using consecutive sampling, the sample will include three patient groups representative of the ICU population who: a) can communicate (able to self-report) and exhibit behaviors, b) cannot communicate but can exhibit behaviors, and c) cannot communicate nor exhibit behaviors. Participants will be observed before, during and 15 minutes after non-nociceptive (i.e., soft touch, cuff inflation) and nociceptive procedures (e.g., chest tube or drain removal, endotracheal suctioning, arterial or intravenous catheter insertion, wound care, bed turning) part of standard care. The NOL will be continuously monitored during all these time points, patients able to self-report will rate their 0-10 pain intensity and procedural pain distress, and patients unable to self-report in whom behaviors are observable will be assessed with the CPOT. Analgesic and sedative agent use will also be documented. Mixed linear models for repeated measures will be used to compare time points, procedures, and their interactions. Receiver Operating Characteristic curve analysis of the NOL will be performed using self-reported pain intensity and CPOT scores as reference criteria. A convenience sample of ICU nurses will also be recruited to offer them the opportunity to learn more about the NOL device, to be exposed to its application at the bedside, and to evaluate its feasibility and potential clinical utility for ICU pain assessment.

The expected outcomes include the validation of a multi-parameter technology in a new context of care which could be used as an alternative measure to detect nociception and related pain and to improve pain management and evaluation of analgesia effectiveness in vulnerable ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU for more than 24 hours
* French or English speaking
* Able to self-report or not
* Negative on delirium screening and not treated for psychosis (patients able to self- report)

Exclusion Criteria:

* Lack an available finger to install the NOL's finger probe
* Suffer severe peripheral vascular disease affecting the upper limbs
* Serious and uncontrolled cardiac arrhythmia
* Are in a hypoperfusion state or shock for which they are receiving high doses of Norepinephrine (>14 mcg/min) or equivalent vasopressors to maintain a SBP >90mmHg or a MAP >65mmHg
* Are agitated (RASS scores from +1 to +4)
* Diagnosed with cognitive deficits (e.g., Alzheimer)
* Are positive for C. Difficile
* Are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive sampling will be used to capture a representative sample of ICU patients able or not to self-report. The study sample will include three ICU patient groups: Group A can communicate using self-report and can exhibit behaviors (conscious and alert with GCS [Glasgow Coma Scale] score of 13 to 15 and RASS [Richmond Agitation Sedation Scale] score of 0), Group B cannot communicate using self-report but can exhibit behaviors (altered level of consciousness with GCS score of 6 to 12 with a score ≥4 on the motor subscale and/or RASS score of -1 to -3), and Group C cannot communicate (GCS 3 to 5) nor exhibit behaviors (unconscious with GCS score of 3 to 5 with a score ≤3 on the motor subscale and RASS score -4 or -5 and/or receiving neuromuscular blocking agents).
Sampling Method: Non-Probability Sample
Enrollment: 411 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Nociception Level Index (NOL) | Before, during soft touch procedure, during cuff inflation procedure, and 15 minutes post
  The Pain Monitoring Device-200 (PMD-200)TM, which offers the multi-parametric NOL index from 0 to 100 (Medasense Biometrics Ltd., Ramat Gan, Israel) will be used. Values >25 were found to be indicative of nociception and related-pain in the field of anesthesia.
Nociception Level Index (NOL) | Before, during a standard care procedure, and 15 minutes post
  The Pain Monitoring Device-200 (PMD-200)TM, which offers the multi-parametric NOL index from 0 to 100 (Medasense Biometrics Ltd., Ramat Gan, Israel) will be used. Values >25 were found to be indicative of nociception and related-pain in the field of anesthesia.
Nociception Level Index (NOL) | Before an opioid dose and 15 minutes post-dose
  The Pain Monitoring Device-200 (PMD-200)TM, which offers the multi-parametric NOL index from 0 to 100 (Medasense Biometrics Ltd., Ramat Gan, Israel) will be used. Values >25 were found to be indicative of nociception and related-pain in the field of anesthesia.

SECONDARY OUTCOMES:
Pain intensity score | Before, during soft touch procedure, during cuff inflation procedure, and 15 minutes post
  The 0-10 Faces Pain Thermometer will be used as a self-report pain intensity scale. It consists of an enlarged visual thermometer including 6 faces with numeric rating scale scoring from 0 "no pain" to 10 "worst possible pain".
Pain intensity score | Before, during a standard care procedure, and 15 minutes post
  The 0-10 Faces Pain Thermometer will be used as a self-report pain intensity scale. It consists of an enlarged visual thermometer including 6 faces with numeric rating scale scoring from 0 "no pain" to 10 "worst possible pain".
Pain intensity score | Before an opioid dose and 15 minutes post-dose
  The 0-10 Faces Pain Thermometer will be used as a self-report pain intensity scale. It consists of an enlarged visual thermometer including 6 faces with numeric rating scale scoring from 0 "no pain" to 10 "worst possible pain".
Behavior pain score | Before, during soft touch procedure, during cuff inflation procedure, and 15 minutes post
  The Critical-Care Pain Observation Tool (CPOT) will be used as a behavioral assessment tool. It includes 4 behavioral domains: 1) facial expressions, 2) body movements, 3) muscle tension, and 4) compliance with the ventilator (for mechanically ventilated patients) or vocalization (for non-intubated patients). Each domain is scored from 0-2, and the total score can range from 0-8. A CPOT score >2 was found to adequately identify patients with pain (as per self-report).
Behavior pain score | Before, during a standard care procedure, and 15 minutes post
  The Critical-Care Pain Observation Tool (CPOT) will be used as a behavioral assessment tool. It includes 4 behavioral domains: 1) facial expressions, 2) body movements, 3) muscle tension, and 4) compliance with the ventilator (for mechanically ventilated patients) or vocalization (for non-intubated patients). Each domain is scored from 0-2, and the total score can range from 0-8. A CPOT score >2 was found to adequately identify patients with pain (as per self-report).
Behavior pain score | Before an opioid dose and 15 minutes post-dose
  The Critical-Care Pain Observation Tool (CPOT) will be used as a behavioral assessment tool. It includes 4 behavioral domains: 1) facial expressions, 2) body movements, 3) muscle tension, and 4) compliance with the ventilator (for mechanically ventilated patients) or vocalization (for non-intubated patients). Each domain is scored from 0-2, and the total score can range from 0-8. A CPOT score >2 was found to adequately identify patients with pain (as per self-report).
Pain distress score | At the end of standard care procedure up to one minute post
  The 0-10 NRS will be used to assess the procedural pain distress experienced by patients during nociceptive procedures. Procedural pain distress is scored on a numeric scale from 0 "not at all distressful" to 10 "most distressful feeling possible".

CONTACTS AND LOCATIONS:
Overall Officials: Céline Gélinas, PhD, RN, Principal Investigator — McGill University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gelinas C, Shahiri T S, Wang HT, Gallani MC, Oulehri W, Laporta D, Richebe P. Validation of the Nociception Level Index for the Detection of Nociception and Pain in Critically Ill Adults: Protocol for an Observational Study. JMIR Res Protoc. 2025 Feb 28;14:e60672. doi: 10.2196/60672. PMID 40053798